CLINICAL TRIAL: NCT02691312
Title: Prevalence and Characterization of Retinopathy in Children With Type 1 Diabetes Using a Non-mydriatic Fundus Camera
Brief Title: Pediatric Type 1 Diabetes and Retinopathy
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201501086
Record Dates: First submitted 2016-02-22; First posted 2016-02-25 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Diabetic Retinopathy
Keywords: type 1 diabetes; retinopathy
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus, Type 1; Retinal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Type 1 diabetes (T1D): Pediatric patients with type 1 diabetes (T1D) will have an eye exam using the Digital Retinography System (DRS) taking non-mydriatic fundus images. If the test is positive or inconclusive, subjects will be notified and referred to an ophthalmologist for a dilated retinal exam. A chart review and questionnaire will be completed to evaluate for risk factors predisposing subjects to diabetic retinopathy.
  Interventions: Device: Digital Retinography System

INTERVENTIONS:
Device: Digital Retinography System — The DRS is a portable non-mydriatic fundus camera in which children place their chin on a chin rest and the camera, after auto-focusing, takes photographs of their retinas. These photographs will be examined by an ophthalmologist (specializing in retinal disease) to assess for evidence of diabetic retinopathy.
  Other Names: CenterVue Digital Retinography System; DRS

SUMMARY:
Diabetic retinopathy (DR) causes more new cases of blindness among young adults than any other disease. More than 90% of individuals with type 1 diabetes (T1D) will have some form of DR by 20 years after their diagnosis. DR is associated with long-term hyperglycemia and blood glucose variability, which induces vascular endothelial dysfunction and destruction in the retina, eventual retinal ischemia, and in the end, widespread neovascularization of the retina and optic disk. When these fragile vessels bleed, they can cause vitreous hemorrhage and loss of vision. Eventually the friable vessels fibrose and can result in retinal detachment or further retinal ischemia.

Major risk factors for the development of diabetic retinopathy are time since diagnosis, age at diagnosis, and severity of hyperglycemia. Retinopathy most commonly occurs at least three years after diagnosis and most cases are diagnosed more than five years after the onset of T1D. Current guidelines from the American Diabetes Association (ADA) and American Academy of Ophthalmology (AAO) recommend that patients with T1D undergo an initial comprehensive dilated fundoscopic evaluation once the individual has had diabetes for 3-5 years and has either reached puberty or 10 years of age, whichever is earlier. These patients should receive a yearly exam thereafter, or every two years based upon the recommendation of an eye care professional. However, the prevalence of retinopathy in children is unknown and adherence to these guidelines, especially in youth, has proven difficult. Thus, it is important to make these guidelines more evidence based, as retinopathy is often asymptomatic until vision loss occurs. The first step in this process is the determination of the prevalence of retinopathy in a general population of youth with diabetes. This should be followed by determining which children are most at risk, so the guidelines can provide realistic and pertinent guidance to practitioners.

DETAILED DESCRIPTION:
The study will be a prospective cross-sectional study of pediatric participants who have had T1D for one year or more. Pediatric participants will be recruited at the Florida Diabetes Camps, the Children With Diabetes Friends for Life Orlando Conference, and the University of Florida Pediatric Endocrinology Clinics. The participants will be tested for diabetic retinopathy using a Digital Retinography System (DRS) (http://www.centervue.com/producta556.html?id=637). The DRS is a portable non-mydriatic fundus camera in which the participants places their chins on the chin-rest and the device takes a digital image of their eyes for evaluation by an ophthalmologist remotely. These photographs will be examined by an ophthalmologist (specializing in retinal disease) to assess for evidence of diabetic retinopathy.

As part of their informed consent, all participants will be asked as part of their informed consent to allow study staff to contact their local ophthalmologist for their eye exam results following a positive or inconclusive portable retinal screening. Participants or their guardians will also be asked to fill out a study questionnaire during the screening visit. When available, the study subjects' medical record will be accessed to identify their BMI, time since T1D diagnosis, previous hemoglobin A1c (HbA1c) levels over the last 12 months (or longer if available), insulin regimen, Tanner staging, serum lipids, urine microalbumin:creatinine, presence or absence of hypertension, and previous diagnoses of diabetic retinopathy, microalbuminuria, hyperlipidemia or hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 diabetes
* Duration of diabetes 1 year or greater

Exclusion Criteria:

* Diabetes less than 1 year duration
* Age < 9 years and >26 years of age

Ages: 9 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: People with type 1 diabetes and a duration of 1 year or greater will be asked to participate. Potential participants will be approached at the Pediatric Endocrinology clinic visits, Florida Diabetes Camp and the Children With Diabetes annual meeting.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-01-20 (Actual); Study Completion 2018-12-27 (Actual)

PRIMARY OUTCOMES:
Number of participants diagnosed with retinopathy | Baseline
  Using a CenterVue Digital Retinography System (DRS) the participants with a positive or inconclusive screen will be called with the results and recommended to undergo a dilated eye examination by a skilled ophthalmologist. The results from the ophthalmologist will be compared to the DRS results.

CONTACTS AND LOCATIONS:
Overall Officials: Janet H Silverstein, MD, Principal Investigator — University of Florida
Locations (3):
- United States (3):
  - Florida Diabetes Camps, De Leon Springs, Florida
  - Pediatrics Endocrinology/Diabetes at UF Health Medical Plaza and Children's Medical Services Building, Gainesville, Florida
  - Children With Diabetes Friends For Life Conference, Orlando, Florida

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- Available data/document: FDA 501(k) — https://www.accessdata.fda.gov/cdrh_docs/pdf10/K101935.pdf